CLINICAL TRIAL: NCT04244838
Title: Biomechanical Functional Evaluation Through Gait Analysis in Patients Underwent Total Knee Arthroplasty With a Medial Pivot Design: Pilot Study
Brief Title: Gait Analysis in Patients Underwent Total Knee Arthroplasty With a Medial Pivot Design.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-TKA-GAIT
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis
Keywords: Medially stabilized total knee arthroplasty; In vivo kinematics; gait analysis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MP-TKA group (Experimental): 20 patients candidates for cemented TKA with MP design for tri-compartment gonarthrosis will be recruited on indications of the surgeon and according to normal clinical practice at the Orthopedic and Traumatological Clinic 2nd of the Rizzoli Orthopedic Institute.
  Interventions: Diagnostic Test: Gait Analysis

INTERVENTIONS:
Diagnostic Test: Gait Analysis — The patients will undergo Gait analysis (integrated movement analysis system) performed at the Complex Laboratory for Movement Analysis and functional-clinical evaluation of the prosthesis of the Rizzoli Orthopedic Institute. The instrumentation used in the Movement Analysis Laboratory consists of a stereophotogrammetric system equipped with eight infrared cameras (Vicon® 460-Oxford system) and 2 dynamometric platforms (Kistler® Instrument, AG Switzerland). The IOR GAIT protocol will be used as a marker set (Leardini et al. 2007). For the evaluation of muscle activation, surface electromyography with 16-channel system will be used (ZeroWire Cometa, Milan). Spatio-temporal parameters, kinematics, kinetics and muscle activation will be evaluated.

SUMMARY:
The purpose of the present pilot study is to evaluate, through gait analysis and rating scales, the functional outcome during the execution of motor tasks with high functional demand such as walking on an unstable surface, stair ascent and descent, maximal knee flexion under load (lunge) on a sample of 20 subjects candidates to cemented total knee arthroplasty with MP design at the Orthopedic and Traumatology Clinic 2nd of the Rizzoli Orthopedic Institute. The parameters obtained will be compared with the parameters of healthy subjects comparable by age and Body Max Index (BMI) already acquired at the Movement Analysis Laboratory of the Rizzoli Orthopedic Institute, where the study will be conducted.

On the day of admission to the ward (generally the day before the scheduled surgery), the enrolled patients will undergo the evaluation scales and gait analysis at the Institute's Movement Analysis Laboratory.

The patients will be operated by the team of the Traumatological Orthopedic Clinic 2nd through the implantation of a cemented total knee prosthesis MP (Evolution medial-pivot knee system, MicroPort Orthopedics). Anterior knee access with medial para-patellar capsulotomy and standard instruments will be used according to current standards of good clinical practice.

In the post-operative period, patients will carry out post-surgical rehabilitation following normal clinical practice.

The patients will be re-evaluated at a 6-month follow-up through gait analysis and evaluation scales on the occasion of the control visit that takes place, according to the normal clinical practice at the Institute.

DETAILED DESCRIPTION:
Total knee prosthesis (PTG) is a widespread surgical procedure that aims to treat severe knee osteoarthritis. This type of intervention has proved successful in reducing chronic pain caused by osteoarthritis and in improving the motor performance of the operated subject as well as the quality of life even if the functional outcome after this procedure is still limited, especially in the execution of more complex and demanding motor tasks (e.g. climbing and descending stairs, walking on unstable surfaces, maximum knee flexion under load) due to the difficulty in finding a prosthetic design that mimics the natural joint biomechanics of a non-arthrosic knee.

Medial Pivot (MP) knee prostheses have been designed to meet these requirements by replicating the morphology of the healthy knee, characterized by a medial compartment with a stable conformation and a movable lateral compartment that moves by rotating around the pivot point. Despite the theoretical premises of this prosthetic model, in literature very few studies have investigated how the MP design translates into an improvement of the functional outcome of the subject operated during the journey, while no study has ever been conducted to evaluate the functional outcome during the execution of more demanding motor tasks although the subjects who undergo knee arthroplasty are always younger and more and more active, with increasingly higher functional needs. To date, gait analysis, a non-invasive functional assessment method that provides objective and quantitative data about spatio-temporal parameters, kinematics, kinetics and muscle activation, represents the Gold Standard for the assessment of functional outcome both in healthy patients and in patients subjected to prosthetic surgery.

The purpose of the present pilot study is to evaluate, through gait analysis and rating scales, the functional outcome during the execution of motor tasks with high functional demand such as walking on an unstable surface, stair ascent and descent, maximal knee flexion under load (lunge) on a sample of 20 subjects candidates to cemented total knee arthroplasty with MP design at the Orthopedic and Traumatology Clinic 2nd of the Rizzoli Orthopedic Institute. The parameters obtained will be compared with the parameters of healthy subjects comparable by age and Body Max Index (BMI) already acquired at the Movement Analysis Laboratory of the Rizzoli Orthopedic Institute, where the study will be conducted.

The pilot study is necessary to carry out a preliminary assessment of the functional outcome and joint biomechanics of the knee prosthesis with the gait analysis method never performed in other studies during the execution of demanding motor tasks, with high functional demand. The collection of information and data obtained will allow the appropriate calculation of the sample useful for a subsequent study.

During the pre-hospitalization visit, participation in the study will be proposed to those who meet the inclusion criteria. If the subject accepts, he will be recruited and will have to sign the informed consent to the study.

On the day of admission to the ward (generally the day before the scheduled surgery), the enrolled patients will undergo the evaluation scales and gait analysis at the Institute's Movement Analysis Laboratory.

The patients will be operated by the team of the Traumatological Orthopedic Clinic 2nd through the implantation of a cemented total knee prosthesis MP (Evolution medial-pivot knee system, MicroPort Orthopedics). Anterior knee access with medial para-patellar capsulotomy and standard instruments will be used according to current standards of good clinical practice.

In the post-operative period, patients will carry out post-surgical rehabilitation following normal clinical practice.

The patients will be re-evaluated at a 6-month follow-up through gait analysis and evaluation scales on the occasion of the control visit that takes place, according to the normal clinical practice at the Institute.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-75 years of both gender
* Patients with three-compartment knee arthrosis (primary or secondary post-traumatic)
* Patients with femoral or tibial osteonecrosis
* Patients with posterior cruciate ligament and healthy collateral ligaments at the level of the affected knee
* Deformity in varus or valgus inferior to 10 °
* Person able to provide informed consent and who agrees to sign the Informed Consent Form approved by the Ethics Committee (EC).
* Subject compliant with post-operative rehabilitation to be performed according to normal clinical practice

Exclusion Criteria:

* Patients with severe morphostructural alterations or other pathologies affecting the knee and lower limb
* Patients with serious systemic vascular and neurological pathologies
* Obese or body mass index BMI> 30 kg / m2
* Patients with posterior cruciate ligament and / or collateral ligaments injury in the affected knee
* Knee arthroplasty in the contralateral
* Patient not compliant with post-operative rehabilitation

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-05-19 (Actual)

PRIMARY OUTCOMES:
Gait analysis | 20 months
  Spatio-temporal parameters, kinematics of pelvis, hip, knee and ankle in the sagittal coronal and transverse planes, kinetics (joint moments and foot-soil reaction forces), rectus femoral muscle activation, biceps femoris, anterior tibialis, medial twin during the path, ascent and descent from stairs, lunge, path on unstable surface
American Knee Society Score | 22 months
  It is used to assess knee functionality by investigator. It consists of both a clinical and a functional score
Knee injury and Osteoarthritis Outcome Score | 22 months
  KOOS is a valid, reliable and responsive self-administered instrument that can be used for short-term and long-term follow-up of several types of knee injury including osteoarthritis.
  It consists of five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QoL).
Visual analogue scale | 22 months
  It is used for subjective pain evaluation
Short Form-36 | 22 months
  36 items presented in eight dimensions (physical activity, monitoring of the role due to physical health, emotional state, physical pain, perception of the general state of health, vitality, social activities and mental health).

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Maria Marcheggiani Muccioli, MD, PhD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alnahdi AH, Zeni JA, Snyder-Mackler L. Gait after unilateral total knee arthroplasty: frontal plane analysis. J Orthop Res. 2011 May;29(5):647-52. doi: 10.1002/jor.21323. Epub 2010 Dec 23. PMID 21437943
- [Result] Benjamin B, Pietrzak JRT, Tahmassebi J, Haddad FS. A functional comparison of medial pivot and condylar knee designs based on patient outcomes and parameters of gait. Bone Joint J. 2018 Jan;100-B(1 Supple A):76-82. doi: 10.1302/0301-620X.100B1.BJJ-2017-0605.R1. PMID 29292344
- [Result] Hatfield GL, Hubley-Kozey CL, Astephen Wilson JL, Dunbar MJ. The effect of total knee arthroplasty on knee joint kinematics and kinetics during gait. J Arthroplasty. 2011 Feb;26(2):309-18. doi: 10.1016/j.arth.2010.03.021. Epub 2010 May 31. PMID 20570095
- [Result] Hubley-Kozey CL, Hatfield GL, Astephen Wilson JL, Dunbar MJ. Alterations in neuromuscular patterns between pre and one-year post-total knee arthroplasty. Clin Biomech (Bristol). 2010 Dec;25(10):995-1002. doi: 10.1016/j.clinbiomech.2010.07.008. Epub 2010 Aug 21. PMID 20728970
- [Result] Leardini A, Sawacha Z, Paolini G, Ingrosso S, Nativo R, Benedetti MG. A new anatomically based protocol for gait analysis in children. Gait Posture. 2007 Oct;26(4):560-71. doi: 10.1016/j.gaitpost.2006.12.018. Epub 2007 Feb 8. PMID 17291764
- [Result] Levinger P, Menz HB, Morrow AD, Perrott MA, Bartlett JR, Feller JA, Bergman NB. Knee biomechanics early after knee replacement surgery predict abnormal gait patterns 12 months postoperatively. J Orthop Res. 2012 Mar;30(3):371-6. doi: 10.1002/jor.21545. Epub 2011 Sep 1. PMID 21887700
- [Result] McIntosh AS, Beatty KT, Dwan LN, Vickers DR. Gait dynamics on an inclined walkway. J Biomech. 2006;39(13):2491-502. doi: 10.1016/j.jbiomech.2005.07.025. Epub 2005 Sep 15. PMID 16169000
- [Result] Moonot P, Mu S, Railton GT, Field RE, Banks SA. Tibiofemoral kinematic analysis of knee flexion for a medial pivot knee. Knee Surg Sports Traumatol Arthrosc. 2009 Aug;17(8):927-34. doi: 10.1007/s00167-009-0777-1. Epub 2009 Mar 31. PMID 19333579
- [Result] Naal FD, Fischer M, Preuss A, Goldhahn J, von Knoch F, Preiss S, Munzinger U, Drobny T. Return to sports and recreational activity after unicompartmental knee arthroplasty. Am J Sports Med. 2007 Oct;35(10):1688-95. doi: 10.1177/0363546507303562. Epub 2007 Jun 8. PMID 17557876